CLINICAL TRIAL: NCT01491178
Title: Post-Marketing Surveillance on the Long-Term Use of Prazaxa® Capsules in Patients With Nonvalvular Atrial Fibrillation
Brief Title: Post-Marketing Surveillance of Prazaxa® on the Long-term Use in Patients With Nonvalvular Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.130
Record Dates: First submitted 2011-12-12; First posted 2011-12-13 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2017-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with NVAF
  Interventions: Drug: Prazaxa

INTERVENTIONS:
Drug: Prazaxa — Dabigatran etexilate

SUMMARY:
To investigate the safety and efficacy of long-term use of Prazaxa® Capsules in patients with nonvalvular atrial fibrillation for preventing the occurrence of ischemic stroke or systemic embolism (SEE).

ELIGIBILITY:
Inclusion criteria:

- Patients with nonvalvular atrial fibrillation who have never received Prazaxa Capsules for preventing the occurrence of ischemic stroke and systemic embolism will be included.

Exclusion criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 5000
Sampling Method: Non-Probability Sample
Enrollment: 6772 (Actual)
Dates: Start 2011-12-12 (Actual); Primary Completion 2016-08-02 (Actual); Study Completion 2016-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1164):
- Japan (1164):
  - Boehringer Ingelheim Investigational Site 1, Abashiri, Hokkaido
  - Boehringer Ingelheim Investigational Site 287, Adachi,Tokyo
  - Boehringer Ingelheim Investigational Site 288, Adachi,Tokyo
  - Boehringer Ingelheim Investigational Site 289, Adachi,Tokyo
  - Boehringer Ingelheim Investigational Site 290, Adachi,Tokyo
  - Boehringer Ingelheim Investigational Site 291, Adachi,Tokyo
  - Boehringer Ingelheim Investigational Site 292, Adachi,Tokyo
  - Boehringer Ingelheim Investigational Site 1141, Aira,Kagoshima
  - Boehringer Ingelheim Investigational Site 622, Aisai,Aichi
  - Boehringer Ingelheim Investigational Site 111, Aizuwakamatsu,Fukushima
  - Boehringer Ingelheim Investigational Site 112, Aizuwakamatsu,Fukushima
  - Boehringer Ingelheim Investigational Site 815, Akashi,Hyogo
  - Boehringer Ingelheim Investigational Site 816, Akashi,Hyogo
  - Boehringer Ingelheim Investigational Site 86, Akita,Akita
  - Boehringer Ingelheim Investigational Site 87, Akita,Akita
  - Boehringer Ingelheim Investigational Site 88, Akita,Akita
  - Boehringer Ingelheim Investigational Site 89, Akita,Akita
  - Boehringer Ingelheim Investigational Site 817, Ako,Hyogo
  - Boehringer Ingelheim Investigational Site 818, Ako,Hyogo
  - Boehringer Ingelheim Investigational Site 1142, Akune,Kagoshima
  - Boehringer Ingelheim Investigational Site 819, Amagasaki,Hyogo
  - Boehringer Ingelheim Investigational Site 820, Amagasaki,Hyogo
  - Boehringer Ingelheim Investigational Site 821, Amagasaki,Hyogo
  - Boehringer Ingelheim Investigational Site 822, Amagasaki,Hyogo
  - Boehringer Ingelheim Investigational Site 823, Amagasaki,Hyogo
  - Boehringer Ingelheim Investigational Site 1084, Amakusa,Kumamoto
  - Boehringer Ingelheim Investigational Site 968, Anan,Tokushima
  - Boehringer Ingelheim Investigational Site 969, Anan,Tokushima
  - Boehringer Ingelheim Investigational Site 623, Anjo,Aichi
  - Boehringer Ingelheim Investigational Site 174, Annaka,Gunma
  - Boehringer Ingelheim Investigational Site 45, Aomori,Aomori
  - Boehringer Ingelheim Investigational Site 46, Aomori,Aomori
  - Boehringer Ingelheim Investigational Site 47, Aomori,Aomori
  - Boehringer Ingelheim Investigational Site 48, Aomori,Aomori
  - Boehringer Ingelheim Investigational Site 293, Arakawa,Tokyo
  - Boehringer Ingelheim Investigational Site 877, Arida,Wakayama
  - Boehringer Ingelheim Investigational Site 244, Asahi,Chiba
  - Boehringer Ingelheim Investigational Site 2, Asahikawa,Hokkaido
  - Boehringer Ingelheim Investigational Site 3, Asahikawa,Hokkaido
  - Boehringer Ingelheim Investigational Site 4, Asahikawa,Hokkaido
  - Boehringer Ingelheim Investigational Site 1013, Asakura,Fukuoka
  - Boehringer Ingelheim Investigational Site 157, Ashikaga,Tochigi
  - Boehringer Ingelheim Investigational Site 423, Asigarakami,Kanagawa
  - Boehringer Ingelheim Investigational Site 424, Asigarakami,Kanagawa
  - Boehringer Ingelheim Investigational Site 595, Atami,Shizuoka
  - Boehringer Ingelheim Investigational Site 552, Azumino,Nagano
  - Boehringer Ingelheim Investigational Site 1109, Beppu,Oita
  - Boehringer Ingelheim Investigational Site 903, Bizen,Okayama
  - Boehringer Ingelheim Investigational Site 1110, Bungotakada,Oita
  - Boehringer Ingelheim Investigational Site 294, Bunkyo,Tokyo
  - Boehringer Ingelheim Investigational Site 295, Bunkyo,Tokyo
  - Boehringer Ingelheim Investigational Site 296, Bunkyo,Tokyo
  - Boehringer Ingelheim Investigational Site 297, Bunkyo,Tokyo
  - Boehringer Ingelheim Investigational Site 298, Bunkyo,Tokyo
  - Boehringer Ingelheim Investigational Site 1014, Buzen,Fukuoka
  - Boehringer Ingelheim Investigational Site 245, Chiba,Chiba
  - Boehringer Ingelheim Investigational Site 246, Chiba,Chiba
  - Boehringer Ingelheim Investigational Site 247, Chiba,Chiba
  - Boehringer Ingelheim Investigational Site 248, Chiba,Chiba
  - Boehringer Ingelheim Investigational Site 249, Chiba,Chiba
  - Boehringer Ingelheim Investigational Site 250, Chiba,Chiba
  - Boehringer Ingelheim Investigational Site 251, Chiba,Chiba
  - Boehringer Ingelheim Investigational Site 425, Chigasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 426, Chigasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 553, Chikuma,Nagano
  - Boehringer Ingelheim Investigational Site 554, Chikuma,Nagano
  - Boehringer Ingelheim Investigational Site 127, Chikusei,Ibaraki
  - Boehringer Ingelheim Investigational Site 1015, Chikushino,Fukuoka
  - Boehringer Ingelheim Investigational Site 624, Chita,Aichi
  - Boehringer Ingelheim Investigational Site 299, Chiyoda,Tokyo
  - Boehringer Ingelheim Investigational Site 300, Chiyoda,Tokyo
  - Boehringer Ingelheim Investigational Site 301, Chofu,Tokyo
  - Boehringer Ingelheim Investigational Site 252, Choshi,Chiba
  - Boehringer Ingelheim Investigational Site 302, Chuo,Tokyo
  - Boehringer Ingelheim Investigational Site 90, Daisen,Akita
  - Boehringer Ingelheim Investigational Site 715, Daito,Osaka
  - Boehringer Ingelheim Investigational Site 716, Daito,Osaka
  - Boehringer Ingelheim Investigational Site 113, Date,Fukushima
  - Boehringer Ingelheim Investigational Site 5, Date,Hokkaido
  - Boehringer Ingelheim Investigational Site 6, Date,Hokkaido
  - Boehringer Ingelheim Investigational Site 7, Ebetsu,Hokkaido
  - Boehringer Ingelheim Investigational Site 8, Ebetsu,Hokkaido
  - Boehringer Ingelheim Investigational Site 427, Ebina,Kanagawa
  - Boehringer Ingelheim Investigational Site 428, Ebina,Kanagawa
  - Boehringer Ingelheim Investigational Site 1130, Ebino,Miyazaki
  - Boehringer Ingelheim Investigational Site 1131, Ebino,Miyazaki
  - Boehringer Ingelheim Investigational Site 531, Echizen,Fukui
  - Boehringer Ingelheim Investigational Site 303, Edogawa,Tokyo
  - Boehringer Ingelheim Investigational Site 304, Edogawa,Tokyo
  - Boehringer Ingelheim Investigational Site 305, Edogawa,Tokyo
  - Boehringer Ingelheim Investigational Site 306, Edogawa,Tokyo
  - Boehringer Ingelheim Investigational Site 307, Edogawa,Tokyo
  - Boehringer Ingelheim Investigational Site 308, Edogawa,Tokyo
  - Boehringer Ingelheim Investigational Site 10, Eniwa,Hokkaido
  - Boehringer Ingelheim Investigational Site 9, Eniwa,Hokkaido
  - Boehringer Ingelheim Investigational Site 309, Fuchu,Tokyo
  - Boehringer Ingelheim Investigational Site 310, Fuchu,Tokyo
  - Boehringer Ingelheim Investigational Site 311, Fuchu,Tokyo
  - Boehringer Ingelheim Investigational Site 312, Fuchu,Tokyo
  - Boehringer Ingelheim Investigational Site 537, Fuefuki,Yamanashi
  - Boehringer Ingelheim Investigational Site 596, Fuji,Shizuoka
  - Boehringer Ingelheim Investigational Site 597, Fujieda,Shizuoka
  - Boehringer Ingelheim Investigational Site 195, Fujimi,Saitama
  - Boehringer Ingelheim Investigational Site 429, Fujisawa,Kanagawa
  - Boehringer Ingelheim Investigational Site 430, Fujisawa,Kanagawa
  - Boehringer Ingelheim Investigational Site 431, Fujisawa,Kanagawa
  - Boehringer Ingelheim Investigational Site 432, Fujisawa,Kanagawa
  - Boehringer Ingelheim Investigational Site 433, Fujisawa,Kanagawa
  - Boehringer Ingelheim Investigational Site 538, Fujiyoshida,Yamanashi
  - Boehringer Ingelheim Investigational Site 539, Fujiyoshida,Yamanashi
  - Boehringer Ingelheim Investigational Site 196, Fukaya,Saitama
  - Boehringer Ingelheim Investigational Site 197, Fukaya,Saitama
  - Boehringer Ingelheim Investigational Site 687, Fukuchiyama,Kyoto
  - Boehringer Ingelheim Investigational Site 688, Fukuchiyama,Kyoto
  - Boehringer Ingelheim Investigational Site 532, Fukui,Fukui
  - Boehringer Ingelheim Investigational Site 533, Fukui,Fukui
  - Boehringer Ingelheim Investigational Site 534, Fukui,Fukui
  - Boehringer Ingelheim Investigational Site 1016, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 1017, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 1018, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 1019, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 1020, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 1021, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 1022, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 1023, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 1024, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 1025, Fukuoka,Fukuoka
  - Boehringer Ingelheim Investigational Site 114, Fukushima,Fukushima
  - Boehringer Ingelheim Investigational Site 115, Fukushima,Fukushima
  - Boehringer Ingelheim Investigational Site 116, Fukushima,Fukushima
  - Boehringer Ingelheim Investigational Site 117, Fukushima,Fukushima
  - Boehringer Ingelheim Investigational Site 920, Fukuyama,Hiroshima
  - Boehringer Ingelheim Investigational Site 921, Fukuyama,Hiroshima
  - Boehringer Ingelheim Investigational Site 922, Fukuyama,Hiroshima
  - Boehringer Ingelheim Investigational Site 923, Fukuyama,Hiroshima
  - Boehringer Ingelheim Investigational Site 924, Fukuyama,Hiroshima
  - Boehringer Ingelheim Investigational Site 253, Funabashi,Chiba
  - Boehringer Ingelheim Investigational Site 313, Fussa,Tokyo
  - Boehringer Ingelheim Investigational Site 254, Futtsu,Chiba
  - Boehringer Ingelheim Investigational Site 577, Fuwa,Gifu
  - Boehringer Ingelheim Investigational Site 625, Gamagori,Aichi
  - Boehringer Ingelheim Investigational Site 578, Gifu,Gifu
  - Boehringer Ingelheim Investigational Site 579, Gifu,Gifu
  - Boehringer Ingelheim Investigational Site 580, Gifu,Gifu
  - Boehringer Ingelheim Investigational Site 581, Gifu,Gifu
  - Boehringer Ingelheim Investigational Site 582, Gifu,Gifu
  - Boehringer Ingelheim Investigational Site 583, Gifu,Gifu
  - Boehringer Ingelheim Investigational Site 584, Gifu,Gifu
  - Boehringer Ingelheim Investigational Site 49, Goshogawara,Aomori
  - Boehringer Ingelheim Investigational Site 1069, Goto,Nagasaki
  - Boehringer Ingelheim Investigational Site 1070, Goto,Nagasaki
  - Boehringer Ingelheim Investigational Site 894, Gotsu,Shimane
  - Boehringer Ingelheim Investigational Site 198, Gyoda,Saitama
  - Boehringer Ingelheim Investigational Site 199, Gyoda,Saitama
  - Boehringer Ingelheim Investigational Site 717, Habikino,Osaka
  - Boehringer Ingelheim Investigational Site 718, Habikino,Osaka
  - Boehringer Ingelheim Investigational Site 719, Habikino,Osaka
  - Boehringer Ingelheim Investigational Site 50, Hachinohe,Aomori
  - Boehringer Ingelheim Investigational Site 314, Hachioji,Tokyo
  - Boehringer Ingelheim Investigational Site 315, Hachioji,Tokyo
  - Boehringer Ingelheim Investigational Site 316, Hachioji,Tokyo
  - Boehringer Ingelheim Investigational Site 317, Hachioji,Tokyo
  - Boehringer Ingelheim Investigational Site 318, Hachioji,Tokyo
  - Boehringer Ingelheim Investigational Site 319, Hachioji,Tokyo
  - Boehringer Ingelheim Investigational Site 434, Hadano,Kanagawa
  - Boehringer Ingelheim Investigational Site 948, Hagi,Yamaguchi
  - Boehringer Ingelheim Investigational Site 11, Hakodate,Hokkaido
  - Boehringer Ingelheim Investigational Site 12, Hakodate,Hokkaido
  - Boehringer Ingelheim Investigational Site 13, Hakodate,Hokkaido
  - Boehringer Ingelheim Investigational Site 519, Hakui,Ishikawa
  - Boehringer Ingelheim Investigational Site 520, Hakusan,Ishikawa
  - Boehringer Ingelheim Investigational Site 895, Hamada,Shimane
  - Boehringer Ingelheim Investigational Site 896, Hamada,Shimane
  - Boehringer Ingelheim Investigational Site 598, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 599, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 600, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 601, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 602, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 603, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 604, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 605, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 606, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 607, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 608, Hamamatsu,Shizuoka
  - Boehringer Ingelheim Investigational Site 57, Hanamaki,Iwate
  - Boehringer Ingelheim Investigational Site 626, Handa,Aichi
  - Boehringer Ingelheim Investigational Site 627, Handa,Aichi
  - Boehringer Ingelheim Investigational Site 628, Handa,Aichi
  - Boehringer Ingelheim Investigational Site 629, Handa,Aichi
  - Boehringer Ingelheim Investigational Site 878, Hashimoto,Wakayama
  - Boehringer Ingelheim Investigational Site 879, Hashimoto,Wakayama
  - Boehringer Ingelheim Investigational Site 1003, Hata,Kochi
  - Boehringer Ingelheim Investigational Site 1111, Hayami,Oita
  - Boehringer Ingelheim Investigational Site 200, Hidaka,Saitama
  - Boehringer Ingelheim Investigational Site 201, Hidaka,Saitama
  - Boehringer Ingelheim Investigational Site 202, Hidaka,Saitama
  - Boehringer Ingelheim Investigational Site 925, Higashihiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 128, Higashiibaraki,Ibaraki
  - Boehringer Ingelheim Investigational Site 129, Higashiibaraki,Ibaraki
  - Boehringer Ingelheim Investigational Site 978, Higashikagawa,Kagawa
  - Boehringer Ingelheim Investigational Site 320, Higashikurume, Tokyo
  - Boehringer Ingelheim Investigational Site 67, Higashimatsusima,Miyagi
  - Boehringer Ingelheim Investigational Site 68, Higashimatsusima,Miyagi
  - Boehringer Ingelheim Investigational Site 69, Higashimatsusima,Miyagi
  - Boehringer Ingelheim Investigational Site 203, Higashimatsuyama,Saitama
  - Boehringer Ingelheim Investigational Site 321, Higashimurayama,Tokyo
  - Boehringer Ingelheim Investigational Site 100, Higashine,Yamagata
  - Boehringer Ingelheim Investigational Site 99, Higashine,Yamagata
  - Boehringer Ingelheim Investigational Site 101, Higashiokitama,Yamagata
  - Boehringer Ingelheim Investigational Site 720, Higashiosaka,Osaka
  - Boehringer Ingelheim Investigational Site 721, Higashiosaka,Osaka
  - Boehringer Ingelheim Investigational Site 1132, Higashiusuki,Miyazaki
  - Boehringer Ingelheim Investigational Site 949, Hikari,Yamaguchi
  - Boehringer Ingelheim Investigational Site 204, Hiki,Saitama
  - Boehringer Ingelheim Investigational Site 679, Hikone,Shiga
  - Boehringer Ingelheim Investigational Site 680, Hikone,Shiga
  - Boehringer Ingelheim Investigational Site 824, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 825, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 826, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 827, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 828, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 829, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 830, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 831, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 832, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 833, Himeji,Hyogo
  - Boehringer Ingelheim Investigational Site 508, Himi,Toyama
  - Boehringer Ingelheim Investigational Site 887, Hino,Tottori
  - Boehringer Ingelheim Investigational Site 722, Hirakata,Osaka
  - Boehringer Ingelheim Investigational Site 723, Hirakata,Osaka
  - Boehringer Ingelheim Investigational Site 724, Hirakata,Osaka
  - Boehringer Ingelheim Investigational Site 435, Hiratsuka,Kanagawa
  - Boehringer Ingelheim Investigational Site 14, Hiroo,Hokkaido
  - Boehringer Ingelheim Investigational Site 51, Hirosaki,Aomori
  - Boehringer Ingelheim Investigational Site 52, Hirosaki,Aomori
  - Boehringer Ingelheim Investigational Site 53, Hirosaki,Aomori
  - Boehringer Ingelheim Investigational Site 54, Hirosaki,Aomori
  - Boehringer Ingelheim Investigational Site 926, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 927, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 928, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 929, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 930, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 931, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 932, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 933, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 934, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 935, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 936, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 937, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 938, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 939, Hiroshima,Hiroshima
  - Boehringer Ingelheim Investigational Site 1112, Hita,Oita
  - Boehringer Ingelheim Investigational Site 130, Hitachinaka,Ibaraki
  - Boehringer Ingelheim Investigational Site 131, Hitachinaka,Ibaraki
  - Boehringer Ingelheim Investigational Site 132, Hitachiota,Ibaraki
  - Boehringer Ingelheim Investigational Site 950, Hofu,Yamaguchi
  - Boehringer Ingelheim Investigational Site 951, Hofu,Yamaguchi
  - Boehringer Ingelheim Investigational Site 1133, Hyuga,Miyazaki
  - Boehringer Ingelheim Investigational Site 725, Ibaraki,Osaka
  - Boehringer Ingelheim Investigational Site 726, Ibaraki,Osaka
  - Boehringer Ingelheim Investigational Site 727, Ibaraki,Osaka
  - Boehringer Ingelheim Investigational Site 585, Ibi,Gifu
  - Boehringer Ingelheim Investigational Site 1143, Ibusuki,Kagoshima
  - Boehringer Ingelheim Investigational Site 1144, Ibusuki,Kagoshima
  - Boehringer Ingelheim Investigational Site 1145, Ibusuki,Kagoshima
  - Boehringer Ingelheim Investigational Site 255, Ichihara,Chiba
  - Boehringer Ingelheim Investigational Site 256, Ichihara,Chiba
  - Boehringer Ingelheim Investigational Site 257, Ichihara,Chiba
  - Boehringer Ingelheim Investigational Site 258, Ichikawa,Chiba
  - Boehringer Ingelheim Investigational Site 259, Ichikawa,Chiba
  - Boehringer Ingelheim Investigational Site 1146, Ichikikushikino,Kagoshima
  - Boehringer Ingelheim Investigational Site 630, Ichinomiya,Aichi
  - Boehringer Ingelheim Investigational Site 631, Ichinomiya,Aichi
  - Boehringer Ingelheim Investigational Site 555, Iida,Nagano
  - Boehringer Ingelheim Investigational Site 556, Iida,Nagano
  - Boehringer Ingelheim Investigational Site 557, Iida,Nagano
  - Boehringer Ingelheim Investigational Site 558, Iida,Nagano
  - Boehringer Ingelheim Investigational Site 1026, Iizuka,Fukuoka
  - Boehringer Ingelheim Investigational Site 728, Ikeda,Osaka
  - Boehringer Ingelheim Investigational Site 729, Ikeda,Osaka
  - Boehringer Ingelheim Investigational Site 730, Ikeda,Osaka
  - Boehringer Ingelheim Investigational Site 731, Ikeda,Osaka
  - Boehringer Ingelheim Investigational Site 732, Ikeda,Osaka
  - Boehringer Ingelheim Investigational Site 870, Ikoma,Nara
  - Boehringer Ingelheim Investigational Site 509, Imizu,Toyama
  - Boehringer Ingelheim Investigational Site 559, Ina,Nagano
  - Boehringer Ingelheim Investigational Site 560, Ina,Nagano
  - Boehringer Ingelheim Investigational Site 322, Inagi,Tokyo
  - Boehringer Ingelheim Investigational Site 632, Inazawa,Aichi
  - Boehringer Ingelheim Investigational Site 633, Inuyama,Aichi
  - Boehringer Ingelheim Investigational Site 260, Inzai,Chiba
  - Boehringer Ingelheim Investigational Site 205, Iruma,Saitama
  - Boehringer Ingelheim Investigational Site 206, Iruma,Saitama
  - Boehringer Ingelheim Investigational Site 1071, Isahaya,Nagasaki
  - Boehringer Ingelheim Investigational Site 671, Ise,Mie
  - Boehringer Ingelheim Investigational Site 436, Isehara,Kanagawa
  - Boehringer Ingelheim Investigational Site 175, Isesaki,Gunma
  - Boehringer Ingelheim Investigational Site 176, Isesaki,Gunma
  - Boehringer Ingelheim Investigational Site 133, Ishoika,Ibaraki
  - Boehringer Ingelheim Investigational Site 323, Itabashi,Tokyo
  - Boehringer Ingelheim Investigational Site 324, Itabashi,Tokyo
  - Boehringer Ingelheim Investigational Site 325, Itabashi,Tokyo
  - Boehringer Ingelheim Investigational Site 326, Itabashi,Tokyo
  - Boehringer Ingelheim Investigational Site 327, Itabashi,Tokyo
  - Boehringer Ingelheim Investigational Site 328, Itabashi,Tokyo
  - Boehringer Ingelheim Investigational Site 834, Itami,Hyogo
  - Boehringer Ingelheim Investigational Site 835, Itami,Hyogo
  - Boehringer Ingelheim Investigational Site 970, Itano,Tokushima
  - Boehringer Ingelheim Investigational Site 486, Itoigawa,Niigata
  - Boehringer Ingelheim Investigational Site 1027, Itoshima,Fukuoka
  - Boehringer Ingelheim Investigational Site 118, Iwaki,Fukushima
  - Boehringer Ingelheim Investigational Site 119, Iwaki,Fukushima
  - Boehringer Ingelheim Investigational Site 952, Iwakuni,Yamaguchi
  - Boehringer Ingelheim Investigational Site 953, Iwakuni,Yamaguchi
  - Boehringer Ingelheim Investigational Site 954, Iwakuni,Yamaguchi
  - Boehringer Ingelheim Investigational Site 634, Iwakura,Aichi
  - Boehringer Ingelheim Investigational Site 70, Iwanuma,Miyagi
  - Boehringer Ingelheim Investigational Site 609, Iwata,Shizuoka
  - Boehringer Ingelheim Investigational Site 610, Izu,Shizuoka
  - Boehringer Ingelheim Investigational Site 1147, Izumi,Kagoshima
  - Boehringer Ingelheim Investigational Site 733, Izumi,Osaka
  - Boehringer Ingelheim Investigational Site 734, Izumisano,Osaka
  - Boehringer Ingelheim Investigational Site 735, Izumisano,Osaka
  - Boehringer Ingelheim Investigational Site 897, Izumo,Shimane
  - Boehringer Ingelheim Investigational Site 898, Izumo,Shimane
  - Boehringer Ingelheim Investigational Site 899, Izumo,Shimane
  - Boehringer Ingelheim Investigational Site 487, Joetsu,Niigata
  - Boehringer Ingelheim Investigational Site 488, Joetsu,Niigata
  - Boehringer Ingelheim Investigational Site 736, Kadoma,Osaka
  - Boehringer Ingelheim Investigational Site 521, Kaga,Ishikawa
  - Boehringer Ingelheim Investigational Site 1148, Kagoshima,Kagoshima
  - Boehringer Ingelheim Investigational Site 1149, Kagoshima,Kagoshima
  - Boehringer Ingelheim Investigational Site 1150, Kagoshima,Kagoshima
  - Boehringer Ingelheim Investigational Site 1151, Kagoshima,Kagoshima
  - Boehringer Ingelheim Investigational Site 522, Kahoku,Ishikawa
  - Boehringer Ingelheim Investigational Site 523, Kahoku,Ishikawa
  - Boehringer Ingelheim Investigational Site 737, Kaizuka,Osaka
  - Boehringer Ingelheim Investigational Site 738, Kaizuka,Osaka
  - Boehringer Ingelheim Investigational Site 586, Kakamigahara,Gifu
  - Boehringer Ingelheim Investigational Site 836, Kakogawa,Hyogo
  - Boehringer Ingelheim Investigational Site 837, Kakogawa,Hyogo
  - Boehringer Ingelheim Investigational Site 838, Kakogawa,Hyogo
  - Boehringer Ingelheim Investigational Site 839, Kakogawa,Hyogo
  - Boehringer Ingelheim Investigational Site 840, Kakogawa,Hyogo
  - Boehringer Ingelheim Investigational Site 1085, Kamiamakusa,Kumamoto
  - Boehringer Ingelheim Investigational Site 561, Kamiina,Nagano
  - Boehringer Ingelheim Investigational Site 562, Kamiminochi, Nagano
  - Boehringer Ingelheim Investigational Site 102, Kaminoyama,Yamagata
  - Boehringer Ingelheim Investigational Site 134, Kamisu,Ibaraki
  - Boehringer Ingelheim Investigational Site 135, Kamisu,Ibaraki
  - Boehringer Ingelheim Investigational Site 136, Kamisu,Ibaraki
  - Boehringer Ingelheim Investigational Site 587, Kamo,Gifu
  - Boehringer Ingelheim Investigational Site 489, Kamo,Niigata
  - Boehringer Ingelheim Investigational Site 611, Kamo,Shizuoka
  - Boehringer Ingelheim Investigational Site 524, Kanazawa,Ishikawa
  - Boehringer Ingelheim Investigational Site 525, Kanazawa,Ishikawa
  - Boehringer Ingelheim Investigational Site 526, Kanazawa,Ishikawa
  - Boehringer Ingelheim Investigational Site 527, Kanazawa,Ishikawa
  - Boehringer Ingelheim Investigational Site 528, Kanazawa,Ishikawa
  - Boehringer Ingelheim Investigational Site 529, Kanazawa,Ishikawa
  - Boehringer Ingelheim Investigational Site 1152, Kanoya,Kagoshima
  - Boehringer Ingelheim Investigational Site 158, Kanuma,Tochigi
  - Boehringer Ingelheim Investigational Site 159, Kanuma,Tochigi
  - Boehringer Ingelheim Investigational Site 635, Kariya,Aichi
  - Boehringer Ingelheim Investigational Site 137, Kasama,Ibaraki
  - Boehringer Ingelheim Investigational Site 904, Kasaoka,Okayama
  - Boehringer Ingelheim Investigational Site 871, Kashihara,Nara
  - Boehringer Ingelheim Investigational Site 138, Kashima,Ibaraki
  - Boehringer Ingelheim Investigational Site 1061, Kashima,Saga
  - Boehringer Ingelheim Investigational Site 261, Kashiwa,Chiba
  - Boehringer Ingelheim Investigational Site 262, Kashiwa,Chiba
  - Boehringer Ingelheim Investigational Site 1028, Kasuga,Fukuoka
  - Boehringer Ingelheim Investigational Site 1029, Kasuga,Fukuoka
  - Boehringer Ingelheim Investigational Site 1030, Kasuga,Fukuoka
  - Boehringer Ingelheim Investigational Site 636, Kasugai,Aichi
  - Boehringer Ingelheim Investigational Site 637, Kasugai,Aichi
  - Boehringer Ingelheim Investigational Site 1031, Kasuya,Fukuoka
  - Boehringer Ingelheim Investigational Site 15, Kato, Hokkaido
  - Boehringer Ingelheim Investigational Site 263, Katori,Chiba
  - Boehringer Ingelheim Investigational Site 329, Katsushika,Tokyo
  - Boehringer Ingelheim Investigational Site 330, Katsushika,Tokyo
  - Boehringer Ingelheim Investigational Site 331, Katsushika,Tokyo
  - Boehringer Ingelheim Investigational Site 332, Katsushika,Tokyo
  - Boehringer Ingelheim Investigational Site 333, Katsushika,Tokyo
  - Boehringer Ingelheim Investigational Site 535, Katsuyama,Fukui
  - Boehringer Ingelheim Investigational Site 71, Katta,Miyagi
  - Boehringer Ingelheim Investigational Site 739, Kawachinagano,Osaka
  - Boehringer Ingelheim Investigational Site 207, Kawagoe,Saitama
  - Boehringer Ingelheim Investigational Site 208, Kawaguchi,Saitama
  - Boehringer Ingelheim Investigational Site 209, Kawaguchi,Saitama
  - Boehringer Ingelheim Investigational Site 210, Kawaguchi,Saitama
  - Boehringer Ingelheim Investigational Site 841, Kawanishi,Hyogo
  - Boehringer Ingelheim Investigational Site 437, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 438, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 439, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 440, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 441, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 442, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 443, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 444, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 445, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 446, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 447, Kawasaki,Kanagawa
  - Boehringer Ingelheim Investigational Site 211, Kazo,Saitama
  - Boehringer Ingelheim Investigational Site 212, Kazo,Saitama
  - Boehringer Ingelheim Investigational Site 1086, Kikuchi,Kumamoto
  - Boehringer Ingelheim Investigational Site 1087, Kikuchi,Kumamoto
  - Boehringer Ingelheim Investigational Site 264, Kimitsu,Chiba
  - Boehringer Ingelheim Investigational Site 1153, Kirishima,Kagoshima
  - Boehringer Ingelheim Investigational Site 740, Kishiwada,Osaka
  - Boehringer Ingelheim Investigational Site 334, Kita,Tokyo
  - Boehringer Ingelheim Investigational Site 335, Kita,Tokyo
  - Boehringer Ingelheim Investigational Site 336, Kita,Tokyo
  - Boehringer Ingelheim Investigational Site 91, Kitaakita, Akita
  - Boehringer Ingelheim Investigational Site 177, Kitagunma,Gunma
  - Boehringer Ingelheim Investigational Site 58, Kitakami,Iwate
  - Boehringer Ingelheim Investigational Site 1032, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1033, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1034, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1035, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1036, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1037, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1038, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1039, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1040, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1041, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1042, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 1043, Kitakyushu,Fukuoka
  - Boehringer Ingelheim Investigational Site 16, Kitami,Hokkaido
  - Boehringer Ingelheim Investigational Site 17, Kitami,Hokkaido
  - Boehringer Ingelheim Investigational Site 540, Kitamori,Yamanashi
  - Boehringer Ingelheim Investigational Site 213, Kitamoto,Saitama
  - Boehringer Ingelheim Investigational Site 214, Kitamoto,Saitama
  - Boehringer Ingelheim Investigational Site 638, Kitanagoya,Aichi
  - Boehringer Ingelheim Investigational Site 689, Kizugawa,Kyoto
  - Boehringer Ingelheim Investigational Site 842, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 843, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 844, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 845, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 846, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 847, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 848, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 849, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 850, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 851, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 852, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 853, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 854, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 855, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 856, Kobe,Hyogo
  - Boehringer Ingelheim Investigational Site 1004, Kochi,Kochi
  - Boehringer Ingelheim Investigational Site 1005, Kochi,Kochi
  - Boehringer Ingelheim Investigational Site 1006, Kochi,Kochi
  - Boehringer Ingelheim Investigational Site 1007, Kochi,Kochi
  - Boehringer Ingelheim Investigational Site 1008, Kochi,Kochi
  - Boehringer Ingelheim Investigational Site 1009, Kochi,Kochi
  - Boehringer Ingelheim Investigational Site 337, Kodaira,Tokyo
  - Boehringer Ingelheim Investigational Site 338, Kodaira,Tokyo
  - Boehringer Ingelheim Investigational Site 541, Kofu,Yamanashi
  - Boehringer Ingelheim Investigational Site 542, Kofu,Yamanashi
  - Boehringer Ingelheim Investigational Site 543, Kofu,Yamanashi
  - Boehringer Ingelheim Investigational Site 544, Kofu,Yamanashi
  - Boehringer Ingelheim Investigational Site 545, Kofu,Yamanashi
  - Boehringer Ingelheim Investigational Site 1044, Koga,Fukuoka
  - Boehringer Ingelheim Investigational Site 1045, Koga,Fukuoka
  - Boehringer Ingelheim Investigational Site 139, Koga,Ibakaraki
  - Boehringer Ingelheim Investigational Site 339, Koganei,Tokyo
  - Boehringer Ingelheim Investigational Site 340, Koganei,Tokyo
  - Boehringer Ingelheim Investigational Site 681, Koka,Shiga
  - Boehringer Ingelheim Investigational Site 341, Kokubunji,Tokyo
  - Boehringer Ingelheim Investigational Site 971, Komatsu,Tokushima
  - Boehringer Ingelheim Investigational Site 639, Konan,Aichi
  - Boehringer Ingelheim Investigational Site 120, Koriyama,Fukushima
  - Boehringer Ingelheim Investigational Site 121, Koriyama,Fukushima
  - Boehringer Ingelheim Investigational Site 215, Koshigaya,Saitama
  - Boehringer Ingelheim Investigational Site 216, Koshigaya,Saitama
  - Boehringer Ingelheim Investigational Site 342, Koto,Tokyo
  - Boehringer Ingelheim Investigational Site 343, Koto,Tokyo
  - Boehringer Ingelheim Investigational Site 344, Koto,Tokyo
  - Boehringer Ingelheim Investigational Site 345, Koto,Tokyo
  - Boehringer Ingelheim Investigational Site 346, Koto,Tokyo
  - Boehringer Ingelheim Investigational Site 347, Koto,Tokyo
  - Boehringer Ingelheim Investigational Site 348, Koto,Tokyo
  - Boehringer Ingelheim Investigational Site 217, Kuki,Saitama
  - Boehringer Ingelheim Investigational Site 218, Kuki,Saitama
  - Boehringer Ingelheim Investigational Site 219, Kumagaya,Saitama
  - Boehringer Ingelheim Investigational Site 220, Kumagaya,Saitama
  - Boehringer Ingelheim Investigational Site 1088, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1089, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1090, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1091, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1092, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1093, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1094, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1095, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1096, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1097, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1098, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1099, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 1100, Kumamoto,Kumamoto
  - Boehringer Ingelheim Investigational Site 905, Kurashiki,Okayama
  - Boehringer Ingelheim Investigational Site 906, Kurashiki,Okayama
  - Boehringer Ingelheim Investigational Site 907, Kurashiki,Okayama
  - Boehringer Ingelheim Investigational Site 908, Kurashiki,Okayama
  - Boehringer Ingelheim Investigational Site 909, Kurashiki,Okayama
  - Boehringer Ingelheim Investigational Site 888, Kurayoshi,Tottori
  - Boehringer Ingelheim Investigational Site 889, Kurayoshi,Tottori
  - Boehringer Ingelheim Investigational Site 940, Kure,Hiroshima
  - Boehringer Ingelheim Investigational Site 941, Kure,Hiroshima
  - Boehringer Ingelheim Investigational Site 942, Kure,Hiroshima
  - Boehringer Ingelheim Investigational Site 72, Kurihara,Miyagi
  - Boehringer Ingelheim Investigational Site 1046, Kurume,Fukuoka
  - Boehringer Ingelheim Investigational Site 1047, Kurume,Fukuoka
  - Boehringer Ingelheim Investigational Site 1048, Kurume,Fukuoka
  - Boehringer Ingelheim Investigational Site 1049, Kurume,Fukuoka
  - Boehringer Ingelheim Investigational Site 1050, Kurume,Fukuoka
  - Boehringer Ingelheim Investigational Site 682, Kusatsu,Shiga
  - Boehringer Ingelheim Investigational Site 18, Kushiro
  - Boehringer Ingelheim Investigational Site 19, Kushiro
  - Boehringer Ingelheim Investigational Site 20, Kushiro
  - Boehringer Ingelheim Investigational Site 21, Kushiro
  - Boehringer Ingelheim Investigational Site 1113, Kusu,Oita
  - Boehringer Ingelheim Investigational Site 690, Kyotanabe,Kyoto
  - Boehringer Ingelheim Investigational Site 691, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 692, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 693, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 694, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 695, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 696, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 697, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 698, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 699, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 700, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 701, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 702, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 703, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 704, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 705, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 706, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 707, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 708, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 709, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 710, Kyoto,Kyoto
  - Boehringer Ingelheim Investigational Site 349, Machida,Tokyo
  - Boehringer Ingelheim Investigational Site 178, Maehashi,Gunma
  - Boehringer Ingelheim Investigational Site 179, Maehashi,Gunma
  - Boehringer Ingelheim Investigational Site 180, Maehashi,Gunma
  - Boehringer Ingelheim Investigational Site 181, Maehashi,Gunma
  - Boehringer Ingelheim Investigational Site 182, Maehashi,Gunma
  - Boehringer Ingelheim Investigational Site 183, Maehashi,Gunma
  - Boehringer Ingelheim Investigational Site 184, Maehashi,Gunma
  - Boehringer Ingelheim Investigational Site 711, Maizuru,Kyoto
  - Boehringer Ingelheim Investigational Site 741, Matsubara,Osaka
  - Boehringer Ingelheim Investigational Site 265, Matsudo,Chiba
  - Boehringer Ingelheim Investigational Site 266, Matsudo,Chiba
  - Boehringer Ingelheim Investigational Site 267, Matsudo,Chiba
  - Boehringer Ingelheim Investigational Site 900, Matsue,Shimane
  - Boehringer Ingelheim Investigational Site 563, Matsumoto,Nagano
  - Boehringer Ingelheim Investigational Site 564, Matsumoto,Nagano
  - Boehringer Ingelheim Investigational Site 565, Matsumoto,Nagano
  - Boehringer Ingelheim Investigational Site 566, Matsumoto,Nagano
  - Boehringer Ingelheim Investigational Site 672, Matsusaka,Mie
  - Boehringer Ingelheim Investigational Site 989, Matsuyama,Ehime
  - Boehringer Ingelheim Investigational Site 990, Matsuyama,Ehime
  - Boehringer Ingelheim Investigational Site 991, Matsuyama,Ehime
  - Boehringer Ingelheim Investigational Site 992, Matsuyama,Ehime
  - Boehringer Ingelheim Investigational Site 350, Meguro,Tokyo
  - Boehringer Ingelheim Investigational Site 351, Meguro,Tokyo
  - Boehringer Ingelheim Investigational Site 352, Meguro,Tokyo
  - Boehringer Ingelheim Investigational Site 353, Meguro,Tokyo
  - Boehringer Ingelheim Investigational Site 354, Meguro,Tokyo
  - Boehringer Ingelheim Investigational Site 355, Meguro,Tokyo
  - Boehringer Ingelheim Investigational Site 356, Meguro,Tokyo
  - Boehringer Ingelheim Investigational Site 185, Midori,Gunma
  - Boehringer Ingelheim Investigational Site 1101, Minamata,Kumamoto
  - Boehringer Ingelheim Investigational Site 1102, Minamata,Kumamoto
  - Boehringer Ingelheim Investigational Site 1103, Minamata,Kumamoto
  - Boehringer Ingelheim Investigational Site 122, Minamiaizu,Fukushima
  - Boehringer Ingelheim Investigational Site 546, Minamikoma,Yamanashi
  - Boehringer Ingelheim Investigational Site 1154, Minamikyushu,Kagoshima
  - Boehringer Ingelheim Investigational Site 357, Minato,Tokyo
  - Boehringer Ingelheim Investigational Site 358, Minato,Tokyo
  - Boehringer Ingelheim Investigational Site 359, Minato,Tokyo
  - Boehringer Ingelheim Investigational Site 360, Minato,Tokyo
  - Boehringer Ingelheim Investigational Site 361, Minato,Tokyo
  - Boehringer Ingelheim Investigational Site 362, Minato,Tokyo
  - Boehringer Ingelheim Investigational Site 955, Mine,Yamaguchi
  - Boehringer Ingelheim Investigational Site 742, Minoh,Osaka
  - Boehringer Ingelheim Investigational Site 743, Minoh,Osaka
  - Boehringer Ingelheim Investigational Site 588, Minokamo,Gifu
  - Boehringer Ingelheim Investigational Site 744, Minoshima,Osaka
  - Boehringer Ingelheim Investigational Site 55, Misawa,Aomori
  - Boehringer Ingelheim Investigational Site 612, Mishima,Shizuoka
  - Boehringer Ingelheim Investigational Site 613, Mishima,Shizuoka
  - Boehringer Ingelheim Investigational Site 857, Mita,Hyogo
  - Boehringer Ingelheim Investigational Site 363, Mitaka,Tokyo
  - Boehringer Ingelheim Investigational Site 364, Mitaka,Tokyo
  - Boehringer Ingelheim Investigational Site 140, Mito,Ibaraki
  - Boehringer Ingelheim Investigational Site 141, Mito,Ibaraki
  - Boehringer Ingelheim Investigational Site 142, Mito,Ibaraki
  - Boehringer Ingelheim Investigational Site 1051, Miyako,Fukuoka
  - Boehringer Ingelheim Investigational Site 1052, Miyako,Fukuoka
  - Boehringer Ingelheim Investigational Site 59, Miyako,Iwate
  - Boehringer Ingelheim Investigational Site 60, Miyako,Iwate
  - Boehringer Ingelheim Investigational Site 1134, Miyakonojo,Miyazaki
  - Boehringer Ingelheim Investigational Site 1135, Miyazaki,Miyazaki
  - Boehringer Ingelheim Investigational Site 1136, Miyazaki,Miyazaki
  - Boehringer Ingelheim Investigational Site 1137, Miyazaki,Miyazaki
  - Boehringer Ingelheim Investigational Site 1138, Miyazaki,Miyazaki
  - Boehringer Ingelheim Investigational Site 943, Miyoshi,Hiroshima
  - Boehringer Ingelheim Investigational Site 268, Mobara,Chiba
  - Boehringer Ingelheim Investigational Site 160, Moka,Tochigi
  - Boehringer Ingelheim Investigational Site 161, Moka,Tochigi
  - Boehringer Ingelheim Investigational Site 745, Moriguchi,Osaka
  - Boehringer Ingelheim Investigational Site 61, Morioka,Iwate
  - Boehringer Ingelheim Investigational Site 62, Morioka,Iwate
  - Boehringer Ingelheim Investigational Site 63, Morioka,Iwate
  - Boehringer Ingelheim Investigational Site 143, Moriya,Ibaraki
  - Boehringer Ingelheim Investigational Site 1053, Munakata,Fukuoka
  - Boehringer Ingelheim Investigational Site 490, Murakami,Niigata
  - Boehringer Ingelheim Investigational Site 1010, Muroto,Kochi
  - Boehringer Ingelheim Investigational Site 365, Musashino,Tokyo
  - Boehringer Ingelheim Investigational Site 56, Mutsu,Aomori
  - Boehringer Ingelheim Investigational Site 491, Myoko,Niigata
  - Boehringer Ingelheim Investigational Site 673, Nabari,Mie
  - Boehringer Ingelheim Investigational Site 683, Nagahama,Shiga
  - Boehringer Ingelheim Investigational Site 103, Nagai,Yamagata
  - Boehringer Ingelheim Investigational Site 567, Nagano,Nagano
  - Boehringer Ingelheim Investigational Site 568, Nagano,Nagano
  - Boehringer Ingelheim Investigational Site 569, Nagano,Nagano
  - Boehringer Ingelheim Investigational Site 492, Nagaoka,Niigata
  - Boehringer Ingelheim Investigational Site 493, Nagaoka,Niigata
  - Boehringer Ingelheim Investigational Site 712, Nagaokakyo,Kyoto
  - Boehringer Ingelheim Investigational Site 1072, Nagasaki,Nagasaki
  - Boehringer Ingelheim Investigational Site 1073, Nagasaki,Nagasaki
  - Boehringer Ingelheim Investigational Site 1074, Nagasaki,Nagasaki
  - Boehringer Ingelheim Investigational Site 1075, Nagasaki,Nagasaki
  - Boehringer Ingelheim Investigational Site 1076, Nagasaki,Nagasaki
  - Boehringer Ingelheim Investigational Site 1077, Nagasaki,Nagasaki
  - Boehringer Ingelheim Investigational Site 1078, Nagasaki,Nagasaki
  - Boehringer Ingelheim Investigational Site 1157, Nago,Okinawa
  - Boehringer Ingelheim Investigational Site 640, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 641, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 642, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 643, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 644, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 645, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 646, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 647, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 648, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 649, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 650, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 651, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 652, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 653, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 654, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 655, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 656, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 657, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 658, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 659, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 660, Nagoya,Aichi
  - Boehringer Ingelheim Investigational Site 1158, Naha,Okinawa
  - Boehringer Ingelheim Investigational Site 1159, Nakagami,Okinawa
  - Boehringer Ingelheim Investigational Site 366, Nakano,Tokyo
  - Boehringer Ingelheim Investigational Site 367, Nakano,Tokyo
  - Boehringer Ingelheim Investigational Site 368, Nakano,Tokyo
  - Boehringer Ingelheim Investigational Site 369, Nakano,Tokyo
  - Boehringer Ingelheim Investigational Site 370, Nakano,Tokyo
  - Boehringer Ingelheim Investigational Site 371, Nakano,Tokyo
  - Boehringer Ingelheim Investigational Site 372, Nakano,Tokyo
  - Boehringer Ingelheim Investigational Site 979, Nakatado,Kagawa
  - Boehringer Ingelheim Investigational Site 980, Nakatado,Kagawa
  - Boehringer Ingelheim Investigational Site 1114, Nakatsu,Oita
  - Boehringer Ingelheim Investigational Site 589, Nakatsugawa,Gifu
  - Boehringer Ingelheim Investigational Site 530, Nanao,Ishikawa
  - Boehringer Ingelheim Investigational Site 1011, Nangoku,Kochi
  - Boehringer Ingelheim Investigational Site 713, Nantan,Kyoto
  - Boehringer Ingelheim Investigational Site 872, Nara,Nara
  - Boehringer Ingelheim Investigational Site 269, Narita,Chiba
  - Boehringer Ingelheim Investigational Site 270, Narita,Chiba
  - Boehringer Ingelheim Investigational Site 972, Naruto,Tokushima
  - Boehringer Ingelheim Investigational Site 162, Nasushiobara,Tochigi
  - Boehringer Ingelheim Investigational Site 163, Nasushiobara,Tochigi
  - Boehringer Ingelheim Investigational Site 373, Nerima,Tokyo
  - Boehringer Ingelheim Investigational Site 374, Nerima,Tokyo
  - Boehringer Ingelheim Investigational Site 375, Nerima,Tokyo
  - Boehringer Ingelheim Investigational Site 376, Nerima,Tokyo
  - Boehringer Ingelheim Investigational Site 746, Neyagawa,Osaka
  - Boehringer Ingelheim Investigational Site 747, Neyagawa,Osaka
  - Boehringer Ingelheim Investigational Site 748, Neyagawa,Osaka
  - Boehringer Ingelheim Investigational Site 123, Nihonmatsu,Fukushima
  - Boehringer Ingelheim Investigational Site 494, Niigata,Niigata
  - Boehringer Ingelheim Investigational Site 495, Niigata,Niigata
  - Boehringer Ingelheim Investigational Site 496, Niigata,Niigata
  - Boehringer Ingelheim Investigational Site 497, Niigata,Niigata
  - Boehringer Ingelheim Investigational Site 498, Niigata,Niigata
  - Boehringer Ingelheim Investigational Site 499, Niigata,Niigata
  - Boehringer Ingelheim Investigational Site 500, Niigata,Niigata
  - Boehringer Ingelheim Investigational Site 501, Niigata,Niigata
  - Boehringer Ingelheim Investigational Site 993, Niihama,Ehime
  - Boehringer Ingelheim Investigational Site 994, Niihama,Ehime
  - Boehringer Ingelheim Investigational Site 995, Niihama,Ehime
  - Boehringer Ingelheim Investigational Site 64, Ninohe,Iwate
  - Boehringer Ingelheim Investigational Site 65, Ninohe,Iwate
  - Boehringer Ingelheim Investigational Site 547, Nirasaki,Yamanashi
  - Boehringer Ingelheim Investigational Site 1062, Nishimatsuura,Saga
  - Boehringer Ingelheim Investigational Site 858, Nishinomiya,Hyogo
  - Boehringer Ingelheim Investigational Site 859, Nishinomiya,Hyogo
  - Boehringer Ingelheim Investigational Site 860, Nishinomiya,Hyogo
  - Boehringer Ingelheim Investigational Site 861, Nishinomiya,Hyogo
  - Boehringer Ingelheim Investigational Site 862, Nishinomiya,Hyogo
  - Boehringer Ingelheim Investigational Site 863, Nishinomiya,Hyogo
  - Boehringer Ingelheim Investigational Site 661, Nishio,Aichi
  - Boehringer Ingelheim Investigational Site 377, Nishitokyo,Tokyo
  - Boehringer Ingelheim Investigational Site 864, Nishiwaki,Hyogo
  - Boehringer Ingelheim Investigational Site 865, Nishiwaki,Hyogo
  - Boehringer Ingelheim Investigational Site 548, Nishiyachiyo,Yamanashi
  - Boehringer Ingelheim Investigational Site 662, Nisshin,Aichi
  - Boehringer Ingelheim Investigational Site 901, Nita,Shimane
  - Boehringer Ingelheim Investigational Site 1139, Nobeoka,Miyazaki
  - Boehringer Ingelheim Investigational Site 1140, Nobeoka,Miyazaki
  - Boehringer Ingelheim Investigational Site 271, Noda,Chiba
  - Boehringer Ingelheim Investigational Site 272, Noda,Chiba
  - Boehringer Ingelheim Investigational Site 92, Noshiro,Akita
  - Boehringer Ingelheim Investigational Site 614, Numazu,Shizuoka
  - Boehringer Ingelheim Investigational Site 615, Numazu,Shizuoka
  - Boehringer Ingelheim Investigational Site 536, Nyu,Fukui
  - Boehringer Ingelheim Investigational Site 22, Obihiro,Hokkaido
  - Boehringer Ingelheim Investigational Site 23, Obihiro,Hokkaido
  - Boehringer Ingelheim Investigational Site 663, Obu,Aichi
  - Boehringer Ingelheim Investigational Site 93, Odate,Akita
  - Boehringer Ingelheim Investigational Site 94, Odate,Akita
  - Boehringer Ingelheim Investigational Site 448, Odawara,Kanagawa
  - Boehringer Ingelheim Investigational Site 449, Odawara,Kanagawa
  - Boehringer Ingelheim Investigational Site 95, Oga,Akita
  - Boehringer Ingelheim Investigational Site 590, Ogaki,Gifu
  - Boehringer Ingelheim Investigational Site 591, Ogaki,Gifu
  - Boehringer Ingelheim Investigational Site 1054, Ogori,Fukuoka
  - Boehringer Ingelheim Investigational Site 902, Ohda,Shimane
  - Boehringer Ingelheim Investigational Site 1115, Oita,Oita
  - Boehringer Ingelheim Investigational Site 1116, Oita,Oita
  - Boehringer Ingelheim Investigational Site 1117, Oita,Oita
  - Boehringer Ingelheim Investigational Site 1118, Oita,Oita
  - Boehringer Ingelheim Investigational Site 1119, Oita,Oita
  - Boehringer Ingelheim Investigational Site 1120, Oita,Oita
  - Boehringer Ingelheim Investigational Site 1121, Oita,Oita
  - Boehringer Ingelheim Investigational Site 1122, Oita,Oita
  - Boehringer Ingelheim Investigational Site 1123, Oita,Oita
  - Boehringer Ingelheim Investigational Site 1124, Oita,Oita
  - Boehringer Ingelheim Investigational Site 502, Ojiya,Niigata
  - Boehringer Ingelheim Investigational Site 1055, Okawa,Fukuoka
  - Boehringer Ingelheim Investigational Site 570, Okaya,Nagano
  - Boehringer Ingelheim Investigational Site 910, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 911, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 912, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 913, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 914, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 915, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 916, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 917, Okayama,Okayama
  - Boehringer Ingelheim Investigational Site 664, Okazaki,Aichi
  - Boehringer Ingelheim Investigational Site 1160, Okinawa,Okinawa
  - Boehringer Ingelheim Investigational Site 1161, Okinawa,Okinawa
  - Boehringer Ingelheim Investigational Site 378, Ome,Tokyo
  - Boehringer Ingelheim Investigational Site 684, Omihachiman,Shiga
  - Boehringer Ingelheim Investigational Site 685, Omihachiman,Shiga
  - Boehringer Ingelheim Investigational Site 1079, Omura,Nagasaki
  - Boehringer Ingelheim Investigational Site 1056, Omuta,Fukuoka
  - Boehringer Ingelheim Investigational Site 1057, Omuta,Fukuoka
  - Boehringer Ingelheim Investigational Site 1058, Onga,Fukuoka
  - Boehringer Ingelheim Investigational Site 1059, Onga,Fukuoka
  - Boehringer Ingelheim Investigational Site 944, Onomichi,Hiroshima
  - Boehringer Ingelheim Investigational Site 945, Onomichi,Hiroshima
  - Boehringer Ingelheim Investigational Site 188, Ora,Gunma
  - Boehringer Ingelheim Investigational Site 189, Ora,Gunma
  - Boehringer Ingelheim Investigational Site 749, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 750, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 751, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 752, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 753, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 754, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 755, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 756, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 757, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 758, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 759, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 760, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 761, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 762, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 763, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 764, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 765, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 766, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 767, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 768, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 769, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 770, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 771, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 772, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 773, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 774, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 775, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 776, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 777, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 778, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 779, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 780, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 781, Osaka,Osaka
  - Boehringer Ingelheim Investigational Site 782, Osakasayama,Osaka
  - Boehringer Ingelheim Investigational Site 1155, Oshima,Kagoshima
  - Boehringer Ingelheim Investigational Site 66, Oshu,Iwate
  - Boehringer Ingelheim Investigational Site 186, Ota,Gunma
  - Boehringer Ingelheim Investigational Site 187, Ota,Gunma
  - Boehringer Ingelheim Investigational Site 379, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 380, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 381, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 382, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 383, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 384, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 385, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 386, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 387, Ota,Tokyo
  - Boehringer Ingelheim Investigational Site 24, Otaru,Hokkaido
  - Boehringer Ingelheim Investigational Site 686, Otsu,Shiga
  - Boehringer Ingelheim Investigational Site 549, Otuki,Yamanashi
  - Boehringer Ingelheim Investigational Site 996, Ozu,Ehime
  - Boehringer Ingelheim Investigational Site 997, Ozu,Ehime
  - Boehringer Ingelheim Investigational Site 25, Rumoi,Hokkaido
  - Boehringer Ingelheim Investigational Site 144, Ryugosaki,Ibaraki
  - Boehringer Ingelheim Investigational Site 1125, Saeki,Oita
  - Boehringer Ingelheim Investigational Site 1126, Saeki,Oita
  - Boehringer Ingelheim Investigational Site 1127, Saeki,Oita
  - Boehringer Ingelheim Investigational Site 1128, Saeki,Oita
  - Boehringer Ingelheim Investigational Site 1063, Saga,Saga
  - Boehringer Ingelheim Investigational Site 1064, Saga,Saga
  - Boehringer Ingelheim Investigational Site 1065, Saga,Saga
  - Boehringer Ingelheim Investigational Site 1066, Saga,Saga
  - Boehringer Ingelheim Investigational Site 104, Sagae,Yamagata
  - Boehringer Ingelheim Investigational Site 450, Sagamihara,Kanagawa
  - Boehringer Ingelheim Investigational Site 451, Sagamihara,Kanagawa
  - Boehringer Ingelheim Investigational Site 452, Sagamihara,Kanagawa
  - Boehringer Ingelheim Investigational Site 453, Sagamihara,Kanagawa
  - Boehringer Ingelheim Investigational Site 454, Sagamihara,Kanagawa
  - Boehringer Ingelheim Investigational Site 998, Saijo, Ehime
  - Boehringer Ingelheim Investigational Site 221, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 222, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 223, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 224, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 225, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 226, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 227, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 228, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 229, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 230, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 231, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 232, Saitama,Saitama
  - Boehringer Ingelheim Investigational Site 233, Sakado,Saitama
  - Boehringer Ingelheim Investigational Site 783, Sakai,Osaka
  - Boehringer Ingelheim Investigational Site 784, Sakai,Osaka
  - Boehringer Ingelheim Investigational Site 785, Sakai,Osaka
  - Boehringer Ingelheim Investigational Site 786, Sakai,Osaka
  - Boehringer Ingelheim Investigational Site 787, Sakai,Osaka
  - Boehringer Ingelheim Investigational Site 788, Sakai,Osaka
  - Boehringer Ingelheim Investigational Site 789, Sakai,Osaka
  - Boehringer Ingelheim Investigational Site 981, Sakaide,Kagawa
  - Boehringer Ingelheim Investigational Site 982, Sakaide,Kagawa
  - Boehringer Ingelheim Investigational Site 105, Sakata
  - Boehringer Ingelheim Investigational Site 571, Saku,Nagano
  - Boehringer Ingelheim Investigational Site 273, Sakura,Chiba
  - Boehringer Ingelheim Investigational Site 164, Sakura,Tochigi
  - Boehringer Ingelheim Investigational Site 503, Sanjo,Niigata
  - Boehringer Ingelheim Investigational Site 165, Sano,Tochigi
  - Boehringer Ingelheim Investigational Site 166, Sano,Tochigi
  - Boehringer Ingelheim Investigational Site 983, Sanuki,Kagawa
  - Boehringer Ingelheim Investigational Site 956, Sanyo-onoda,Yamaguchi
  - Boehringer Ingelheim Investigational Site 26, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 27, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 28, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 29, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 30, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 31, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 32, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 33, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 34, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 35, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 36, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 37, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 38, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 39, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 40, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 41, Sapporo,Hokkaido
  - Boehringer Ingelheim Investigational Site 1080, Sasebo,Nagasaki
  - Boehringer Ingelheim Investigational Site 1081, Sasebo,Nagasaki
  - Boehringer Ingelheim Investigational Site 145, Sashima,Ibaraki
  - Boehringer Ingelheim Investigational Site 146, Sashima,Ibaraki
  - Boehringer Ingelheim Investigational Site 234, Sayama,Saitama
  - Boehringer Ingelheim Investigational Site 73, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 74, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 75, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 76, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 77, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 78, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 79, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 80, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 81, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 82, Sendai,Miyagi
  - Boehringer Ingelheim Investigational Site 388, Setagaya,Tokyo
  - Boehringer Ingelheim Investigational Site 389, Setagaya,Tokyo
  - Boehringer Ingelheim Investigational Site 390, Setagaya,Tokyo
  - Boehringer Ingelheim Investigational Site 391, Setagaya,Tokyo
  - Boehringer Ingelheim Investigational Site 392, Setagaya,Tokyo
  - Boehringer Ingelheim Investigational Site 393, Setagaya,Tokyo
  - Boehringer Ingelheim Investigational Site 83, Shibata,Miyagi
  - Boehringer Ingelheim Investigational Site 504, Shibata,Niigata
  - Boehringer Ingelheim Investigational Site 505, Shibata,Niigata
  - Boehringer Ingelheim Investigational Site 190, Shibukawa,Gunma
  - Boehringer Ingelheim Investigational Site 191, Shibukawa,Gunma
  - Boehringer Ingelheim Investigational Site 394, Shibuya,Tokyo
  - Boehringer Ingelheim Investigational Site 1082, Shimabara,Nagasaki
  - Boehringer Ingelheim Investigational Site 616, Shimada,Shizuoka
  - Boehringer Ingelheim Investigational Site 957, Shimonoseki,Yamaguchi
  - Boehringer Ingelheim Investigational Site 958, Shimonoseki,Yamaguchi
  - Boehringer Ingelheim Investigational Site 959, Shimonoseki,Yamaguchi
  - Boehringer Ingelheim Investigational Site 960, Shimonoseki,Yamaguchi
  - Boehringer Ingelheim Investigational Site 395, Shinagawa,Tokyo
  - Boehringer Ingelheim Investigational Site 396, Shinagawa,Tokyo
  - Boehringer Ingelheim Investigational Site 397, Shinagawa,Tokyo
  - Boehringer Ingelheim Investigational Site 880, Shingu,Wakayama
  - Boehringer Ingelheim Investigational Site 398, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 399, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 400, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 401, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 402, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 403, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 404, Shinjuku,Tokyo
  - Boehringer Ingelheim Investigational Site 572, Shiojiri,Nagano
  - Boehringer Ingelheim Investigational Site 124, Shirakawa,Fukushima
  - Boehringer Ingelheim Investigational Site 125, Shirakawa,Fukushima
  - Boehringer Ingelheim Investigational Site 274, Shiroi,Chiba
  - Boehringer Ingelheim Investigational Site 84, Shiroishi,Miyagi
  - Boehringer Ingelheim Investigational Site 85, Shiroishi,Miyagi
  - Boehringer Ingelheim Investigational Site 617, Shizuoka,Shizuoka
  - Boehringer Ingelheim Investigational Site 618, Shizuoka,Shizuoka
  - Boehringer Ingelheim Investigational Site 619, Shizuoka,Shizuoka
  - Boehringer Ingelheim Investigational Site 620, Shizuoka,Shizuoka
  - Boehringer Ingelheim Investigational Site 621, Shizuoka,Shizuoka
  - Boehringer Ingelheim Investigational Site 946, Shobara,Hiroshima
  - Boehringer Ingelheim Investigational Site 961, Shunan,Yamaguchi
  - Boehringer Ingelheim Investigational Site 962, Shunan,Yamaguchi
  - Boehringer Ingelheim Investigational Site 235, Soka,Saitama
  - Boehringer Ingelheim Investigational Site 236, Soka,Saitama
  - Boehringer Ingelheim Investigational Site 237, Soka,Saitama
  - Boehringer Ingelheim Investigational Site 238, Soka,Saitama
  - Boehringer Ingelheim Investigational Site 239, Soka,Saitama
  - Boehringer Ingelheim Investigational Site 275, Sosa,Chiba
  - Boehringer Ingelheim Investigational Site 276, Sosa,Chiba
  - Boehringer Ingelheim Investigational Site 405, Suginami,Tokyo
  - Boehringer Ingelheim Investigational Site 406, Suginami,Tokyo
  - Boehringer Ingelheim Investigational Site 407, Suginami,Tokyo
  - Boehringer Ingelheim Investigational Site 408, Suginami,Tokyo
  - Boehringer Ingelheim Investigational Site 409, Suginami,Tokyo
  - Boehringer Ingelheim Investigational Site 410, Suginami,Tokyo
  - Boehringer Ingelheim Investigational Site 790, Suita,Osaka
  - Boehringer Ingelheim Investigational Site 791, Suita,Osaka
  - Boehringer Ingelheim Investigational Site 792, Suita,Osaka
  - Boehringer Ingelheim Investigational Site 793, Suita,Osaka
  - Boehringer Ingelheim Investigational Site 794, Suita,Osaka
  - Boehringer Ingelheim Investigational Site 795, Suita,Osaka
  - Boehringer Ingelheim Investigational Site 796, Suita,Osaka
  - Boehringer Ingelheim Investigational Site 797, Suita,Osaka
  - Boehringer Ingelheim Investigational Site 126, Sukagawa,Fukushima
  - Boehringer Ingelheim Investigational Site 411, Sumida,Tokyo
  - Boehringer Ingelheim Investigational Site 412, Sumida,Tokyo
  - Boehringer Ingelheim Investigational Site 413, Sumida,Tokyo
  - Boehringer Ingelheim Investigational Site 866, Sumoto,Hyogo
  - Boehringer Ingelheim Investigational Site 1012, Susaki,Kochi
  - Boehringer Ingelheim Investigational Site 573, Suwa,Nagano
  - Boehringer Ingelheim Investigational Site 574, Suwa,Nagano
  - Boehringer Ingelheim Investigational Site 575, Suzaka,Nagano
  - Boehringer Ingelheim Investigational Site 674, Suzuka,Mie
  - Boehringer Ingelheim Investigational Site 414, Tachikawa,Tokyo
  - Boehringer Ingelheim Investigational Site 415, Tachikawa,Tokyo
  - Boehringer Ingelheim Investigational Site 416, Tachikawa,Tokyo
  - Boehringer Ingelheim Investigational Site 592, Tajimi,Gifu
  - Boehringer Ingelheim Investigational Site 918, Takahashi,Okayama
  - Boehringer Ingelheim Investigational Site 984, Takamatsu,Kagawa
  - Boehringer Ingelheim Investigational Site 985, Takamatsu,Kagawa
  - Boehringer Ingelheim Investigational Site 986, Takamatsu,Kagawa
  - Boehringer Ingelheim Investigational Site 987, Takamatsu,Kagawa
  - Boehringer Ingelheim Investigational Site 988, Takamatsu,Kagawa
  - Boehringer Ingelheim Investigational Site 510, Takaoka,Toyama
  - Boehringer Ingelheim Investigational Site 511, Takaoka,Toyama
  - Boehringer Ingelheim Investigational Site 512, Takaoka,Toyama
  - Boehringer Ingelheim Investigational Site 867, Takarazuka,Hyogo
  - Boehringer Ingelheim Investigational Site 192, Takasaki,Gunma
  - Boehringer Ingelheim Investigational Site 193, Takasaki,Gunma
  - Boehringer Ingelheim Investigational Site 798, Takatsuki,Osaka
  - Boehringer Ingelheim Investigational Site 799, Takatsuki,Osaka
  - Boehringer Ingelheim Investigational Site 800, Takatsuki,Osaka
  - Boehringer Ingelheim Investigational Site 801, Takatsuki,Osaka
  - Boehringer Ingelheim Investigational Site 593, Takayama,Gifu
  - Boehringer Ingelheim Investigational Site 947, Takehara,Hiroshima
  - Boehringer Ingelheim Investigational Site 1067, Takeo,Saga
  - Boehringer Ingelheim Investigational Site 675, Taki,Mie
  - Boehringer Ingelheim Investigational Site 1068, Taku,Saga
  - Boehringer Ingelheim Investigational Site 417, Tama,Tokyo
  - Boehringer Ingelheim Investigational Site 418, Tama,Tokyo
  - Boehringer Ingelheim Investigational Site 1104, Tamana,Kumamoto
  - Boehringer Ingelheim Investigational Site 1105, Tamana,Kumamoto
  - Boehringer Ingelheim Investigational Site 881, Tanabe,Wakayama
  - Boehringer Ingelheim Investigational Site 1156, Tarumi,Kagoshima
  - Boehringer Ingelheim Investigational Site 277, Tateyama,Chiba
  - Boehringer Ingelheim Investigational Site 868, Tatsuno,Hyogo
  - Boehringer Ingelheim Investigational Site 873, Tenri,Nara
  - Boehringer Ingelheim Investigational Site 167, Tochigi,Tochigi
  - Boehringer Ingelheim Investigational Site 168, Tochigi,Tochigi
  - Boehringer Ingelheim Investigational Site 240, Toda,Saitama
  - Boehringer Ingelheim Investigational Site 241, Toda,Saitama
  - Boehringer Ingelheim Investigational Site 506, Tokamachi,Niigata
  - Boehringer Ingelheim Investigational Site 242, Tokorozawa,Saitama
  - Boehringer Ingelheim Investigational Site 243, Tokorozawa,Saitama
  - Boehringer Ingelheim Investigational Site 973, Tokushima,Tokushima
  - Boehringer Ingelheim Investigational Site 974, Tokushima,Tokushima
  - Boehringer Ingelheim Investigational Site 975, Tokushima,Tokushima
  - Boehringer Ingelheim Investigational Site 976, Tokushima,Tokushima
  - Boehringer Ingelheim Investigational Site 977, Tokushima,Tokushima
  - Boehringer Ingelheim Investigational Site 42, Tomakomai,Hokkaido
  - Boehringer Ingelheim Investigational Site 43, Tomakomai,Hokkaido
  - Boehringer Ingelheim Investigational Site 1162, Tomigusuku,Okinawa
  - Boehringer Ingelheim Investigational Site 194, Tomioka,Gunma
  - Boehringer Ingelheim Investigational Site 513, Tonami, Tonyama
  - Boehringer Ingelheim Investigational Site 802, Tondabayashi,Osaka
  - Boehringer Ingelheim Investigational Site 999, Toon,Ehime
  - Boehringer Ingelheim Investigational Site 147, Toride,Ibaraki
  - Boehringer Ingelheim Investigational Site 419, Toshima,Tokyo
  - Boehringer Ingelheim Investigational Site 420, Toshima,Tokyo
  - Boehringer Ingelheim Investigational Site 421, Toshima,Tokyo
  - Boehringer Ingelheim Investigational Site 422, Toshima,Tokyo
  - Boehringer Ingelheim Investigational Site 890, Tottori,Tottori
  - Boehringer Ingelheim Investigational Site 891, Tottori,Tottori
  - Boehringer Ingelheim Investigational Site 514, Toyama,Toyama
  - Boehringer Ingelheim Investigational Site 515, Toyama,Toyama
  - Boehringer Ingelheim Investigational Site 516, Toyama,Toyama
  - Boehringer Ingelheim Investigational Site 517, Toyama,Toyama
  - Boehringer Ingelheim Investigational Site 518, Toyama,Toyama
  - Boehringer Ingelheim Investigational Site 665, Toyohashi,Aichi
  - Boehringer Ingelheim Investigational Site 666, Toyohashi,Aichi
  - Boehringer Ingelheim Investigational Site 667, Toyokawa,Aichi
  - Boehringer Ingelheim Investigational Site 803, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 804, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 805, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 806, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 807, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 808, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 809, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 810, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 811, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 812, Toyonaka,Osaka
  - Boehringer Ingelheim Investigational Site 869, Toyooka,Hyogo
  - Boehringer Ingelheim Investigational Site 668, Toyota,Aichi
  - Boehringer Ingelheim Investigational Site 669, Toyota,Aichi
  - Boehringer Ingelheim Investigational Site 676, Tsu,Mie
  - Boehringer Ingelheim Investigational Site 507, Tsubame,Niigata
  - Boehringer Ingelheim Investigational Site 44, Tsubetu, Hokkaido
  - Boehringer Ingelheim Investigational Site 148, Tsuchiura,Ibaraki
  - Boehringer Ingelheim Investigational Site 149, Tsuchiura,Ibaraki
  - Boehringer Ingelheim Investigational Site 150, Tsuchiura,Ibaraki
  - Boehringer Ingelheim Investigational Site 151, Tsukuba,Ibaraki
  - Boehringer Ingelheim Investigational Site 152, Tsukuba,Ibaraki
  - Boehringer Ingelheim Investigational Site 153, Tsukuba,Ibaraki
  - Boehringer Ingelheim Investigational Site 106, Tsuruoka,Yamagata
  - Boehringer Ingelheim Investigational Site 107, Tsuruoka,Yamagata
  - Boehringer Ingelheim Investigational Site 1083, Tsushima,Nagasaki
  - Boehringer Ingelheim Investigational Site 919, Tsuyama,Okayama
  - Boehringer Ingelheim Investigational Site 963, Ube,Yamaguchi
  - Boehringer Ingelheim Investigational Site 964, Ube,Yamaguchi
  - Boehringer Ingelheim Investigational Site 874, Uda,Nara
  - Boehringer Ingelheim Investigational Site 576, Ueda,Nagano
  - Boehringer Ingelheim Investigational Site 714, Uji,Kyoto
  - Boehringer Ingelheim Investigational Site 278, Urayasu,Chiba
  - Boehringer Ingelheim Investigational Site 279, Urayasu,Chiba
  - Boehringer Ingelheim Investigational Site 1163, Urazoe,Okinawa
  - Boehringer Ingelheim Investigational Site 1164, Urazoe,Okinawa
  - Boehringer Ingelheim Investigational Site 154, Ushiku,Ibaraki
  - Boehringer Ingelheim Investigational Site 1129, Usuki,Oita
  - Boehringer Ingelheim Investigational Site 169, Utsunomiya,Tochigi
  - Boehringer Ingelheim Investigational Site 170, Utsunomiya,Tochigi
  - Boehringer Ingelheim Investigational Site 171, Utsunomiya,Tochigi
  - Boehringer Ingelheim Investigational Site 172, Utsunomiya,Tochigi
  - Boehringer Ingelheim Investigational Site 1000, Uwajima, Ehime
  - Boehringer Ingelheim Investigational Site 882, Wakayama,Wakayama
  - Boehringer Ingelheim Investigational Site 883, Wakayama,Wakayama
  - Boehringer Ingelheim Investigational Site 884, Wakayama,Wakayama
  - Boehringer Ingelheim Investigational Site 885, Wakayama,Wakayama
  - Boehringer Ingelheim Investigational Site 886, Wakayama,Wakayama
  - Boehringer Ingelheim Investigational Site 280, Yachimata,Chiba
  - Boehringer Ingelheim Investigational Site 281, Yachimata,Chiba
  - Boehringer Ingelheim Investigational Site 282, Yachiyo,Chiba
  - Boehringer Ingelheim Investigational Site 283, Yachiyo,Chiba
  - Boehringer Ingelheim Investigational Site 284, Yachiyo,Chiba
  - Boehringer Ingelheim Investigational Site 285, Yachiyo,Chiba
  - Boehringer Ingelheim Investigational Site 173, Yaita,Tochigi
  - Boehringer Ingelheim Investigational Site 1106, Yamaga,Kumamoto
  - Boehringer Ingelheim Investigational Site 594, Yamagata,Gifu
  - Boehringer Ingelheim Investigational Site 108, Yamagata,Yamagata
  - Boehringer Ingelheim Investigational Site 109, Yamagata,Yamagata
  - Boehringer Ingelheim Investigational Site 965, Yamaguchi,Yamaguchi
  - Boehringer Ingelheim Investigational Site 966, Yamaguchi,Yamaguchi
  - Boehringer Ingelheim Investigational Site 550, Yamanashi,Yamanashi
  - Boehringer Ingelheim Investigational Site 551, Yamanashi,Yamanashi
  - Boehringer Ingelheim Investigational Site 455, Yamato,Kanagawa
  - Boehringer Ingelheim Investigational Site 875, Yamatokoriyama,Nara
  - Boehringer Ingelheim Investigational Site 876, Yamatotakada,Nara
  - Boehringer Ingelheim Investigational Site 1060, Yame,Fukuoka
  - Boehringer Ingelheim Investigational Site 967, Yanai,Yamaguchi
  - Boehringer Ingelheim Investigational Site 813, Yao,Osaka
  - Boehringer Ingelheim Investigational Site 814, Yao,Osaka
  - Boehringer Ingelheim Investigational Site 670, Yatomi,Aichi
  - Boehringer Ingelheim Investigational Site 1107, Yatsushiro,Kumamoto
  - Boehringer Ingelheim Investigational Site 1108, Yatsushiro,Kumamoto
  - Boehringer Ingelheim Investigational Site 1001, Yawatahama,Ehime
  - Boehringer Ingelheim Investigational Site 1002, Yawatahama,Ehime
  - Boehringer Ingelheim Investigational Site 677, Yokkaichi,Mie
  - Boehringer Ingelheim Investigational Site 678, Yokkaichi,Mie
  - Boehringer Ingelheim Investigational Site 456, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 457, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 458, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 459, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 460, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 461, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 462, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 463, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 464, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 465, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 466, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 467, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 468, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 469, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 470, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 471, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 472, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 473, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 474, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 475, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 476, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 477, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 478, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 479, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 480, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 481, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 482, Yokohama, Kanagawa
  - Boehringer Ingelheim Investigational Site 483, Yokosuka,Kanagawa
  - Boehringer Ingelheim Investigational Site 484, Yokosuka,Kanagawa
  - Boehringer Ingelheim Investigational Site 485, Yokosuka,Kanagawa
  - Boehringer Ingelheim Investigational Site 96, Yokote,Akita
  - Boehringer Ingelheim Investigational Site 97, Yokote,Akita
  - Boehringer Ingelheim Investigational Site 892, Yonago,Tottori
  - Boehringer Ingelheim Investigational Site 893, Yonago,Tottori
  - Boehringer Ingelheim Investigational Site 110, Yonezawa,Yamagata
  - Boehringer Ingelheim Investigational Site 286, Yotsukaido,Chiba
  - Boehringer Ingelheim Investigational Site 155, Yuki,Ibaraki
  - Boehringer Ingelheim Investigational Site 156, Yuki,Ibaraki
  - Boehringer Ingelheim Investigational Site 98, Yuzawa,Akita

REFERENCES:
- [Derived] Koretsune Y, Kusakawa K, Harada KH, Koizumi A, Uchiyama S, Atarashi H, Okumura K, Yasaka M, Yamashita T, Taniguchi A, Fukaya T, Inoue H; for J-dabigatran surveillance and JAPAF study investigators. Characteristics of Japanese Patients with Nonvalvular Atrial Fibrillation on Anticoagulant Treatment: A Descriptive Analysis of J-dabigatran Surveillance and JAPAF Study. Cardiol Ther. 2019 Jun;8(1):43-54. doi: 10.1007/s40119-019-0129-2. Epub 2019 Feb 11. PMID 30746608
- [Derived] Inoue H, Uchiyama S, Atarashi H, Okumura K, Koretsune Y, Yasaka M, Yamashita T, Ohnishi M, Yagi N, Fukaya T; J-Dabigatran Surveillance Investigators. Post-marketing surveillance on the long-term use of dabigatran in Japanese patients with nonvalvular atrial fibrillation: Preliminary report of the J-dabigatran surveillance. J Arrhythm. 2016 Apr;32(2):145-50. doi: 10.1016/j.joa.2015.11.008. Epub 2016 Jan 16. PMID 27092197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Post-Marketing Surveillance on the Long-Term Use of Prazaxa® Capsules in patients with nonvalvular atrial fibrillation
Pre-assignment Details: 6772 subjects were enrolled. Among them, Electronic Case Report Form (eCRF) was not collected for 144 subjects and 185 subjects were excluded because of them not following registration rule, no actual visit or previous treatment experience with Prazaxa, leaving 6443 subjects eligible for study who were enrolled and included in the final study.
Groups:
- Patients With NVAF: Patients with nonvalvular atrial fibrillation (NVAF) taking daily oral dose of Prazaxa® Capsules (Dabigatran etexilate). Dosage of Dabigatran etexilate approved in Japan: 300 milligram (mg) daily (150 mg [as 2 capsules of 75 mg] twice a day (b.i.d)) or 220 mg (110 mg [as 1 capsule of 110 mg] b.i.d)
Period: Overall Study
Arm/Group | Patients With NVAF
Started | 6443 (Started are the enrolled subjects who followed registration rule and for who eCRF was collected.)
Completed | 3649 (Completed is defined as 104 weeks follow-up after enrollment.)
Not Completed | 2794
Not completed — Adverse Event | 1016
Not completed — Improvement of NVAF | 210
Not completed — To conduct invasive treatment | 59
Not completed — Lost to follow-up (unknown reason) | 287
Not completed — Lost to follow-up (changing hospital) | 545
Not completed — To take a contraindication | 20
Not completed — Other than specified above | 657

BASELINE CHARACTERISTICS:
Population: Safety set: This patient set includes all patients who received treatment of Prazaxa® Capsules except those who were found not following registration rule, no actual visit, previous treatment experience with Prazaxa.
Arm/Group | Patients With NVAF
Number analyzed (Participants) | 6443
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2133
  Male | 4310

OUTCOME MEASURES:

1. Primary Outcome: Frequency (Percentage) of Participants With Adverse Drug Reactions
Description: Percentage of participants with adverse drug reactions (ADRs) is presented. An ADR is defined as an adverse event (AE) for which either the investigator or the sponsor (or both) assess the causal relationship to Prazaxa® Capsules either as "Related", "Probably related", or "Cannot be denied".
Time Frame: Up to 104 weeks from first administration of study drug
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Patients With NVAF
Number analyzed (Participants) | 6443
Percentage of participants | 28.2

2. Secondary Outcome: Incidences of Stroke and Systemic Embolism (SEE)
Description: Incidence rate of Stroke and SEE (number of patients per 100 patient year) with 95% confidence interval (CI) is reported. Stroke and SEE were recorded as adverse events (AEs) of special interest. Exact Poisson confidence intervals are presented for incidence rate.
Time Frame: Up to 104 weeks from first administration of study drug
Population: Effectiveness set: This analysis set included all patients who received treatment of Prazaxa® Capsules except those who were found not following registration rule, no actual visit, previous treatment experience with Prazaxa, contraindication and / or who did not suffer from NVAF.
Measure: Number (95% Confidence Interval); unit: Number of patients per 100 patient year
Arm/Group | Patients With NVAF
Number analyzed (Participants) | 6395
Number of patients per 100 patient year | 1.27 [1.04 to 1.54]

ADVERSE EVENTS:
Time Frame: Up to 104 weeks from first administration of study drug
Description: Safety set: This patient set includes all patients who received treatment of Prazaxa® Capsules except those who were found not following registration rule, no actual visit, previous treatment experience with Prazaxa.
Arm/Group | Patients With NVAF
Serious Adverse Events (participants affected / at risk) | 618/6443
Other Adverse Events (participants affected / at risk) | 408/6443
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With NVAF (N=6443)
Pneumonia bacterial (Infections and infestations) | 16
Pneumonia (Infections and infestations) | 13
Cellulitis (Infections and infestations) | 4
Sepsis (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 3
Appendicitis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Osteomyelitis (Infections and infestations) | 2
Pulmonary tuberculosis (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Arteriovenous graft site infection (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Fungal peritonitis (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 6
Pancytopenia (Blood and lymphatic system disorders) | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Marasmus (Metabolism and nutrition disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Cachexia (Metabolism and nutrition disorders) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Feeding disorder (Metabolism and nutrition disorders) | 1
Schizophrenia (Psychiatric disorders) | 4
Delirium (Psychiatric disorders) | 1
Cerebral infarction (Nervous system disorders) | 53
Embolic stroke (Nervous system disorders) | 14
Dementia (Nervous system disorders) | 10
Transient ischaemic attack (Nervous system disorders) | 7
Cerebral haemorrhage (Nervous system disorders) | 5
Epilepsy (Nervous system disorders) | 5
Lacunar infarction (Nervous system disorders) | 5
Cerebellar infarction (Nervous system disorders) | 4
Seizure (Nervous system disorders) | 4
Dementia Alzheimer's type (Nervous system disorders) | 2
Haemorrhage intracranial (Nervous system disorders) | 2
Loss of consciousness (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Ischaemic cerebral infarction (Nervous system disorders) | 2
Thrombotic cerebral infarction (Nervous system disorders) | 2
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2
Brain stem infarction (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral thrombosis (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dyslalia (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
IIIrd nerve paralysis (Nervous system disorders) | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Subdural hygroma (Nervous system disorders) | 1
Miller Fisher syndrome (Nervous system disorders) | 1
Clonic convulsion (Nervous system disorders) | 1
Embolic cerebral infarction (Nervous system disorders) | 1
Cataract (Eye disorders) | 2
Retinal detachment (Eye disorders) | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1
Cardiac failure (Cardiac disorders) | 73
Cardiac failure congestive (Cardiac disorders) | 24
Atrial fibrillation (Cardiac disorders) | 20
Sinus node dysfunction (Cardiac disorders) | 9
Acute myocardial infarction (Cardiac disorders) | 8
Angina pectoris (Cardiac disorders) | 7
Cardiac failure chronic (Cardiac disorders) | 5
Angina unstable (Cardiac disorders) | 4
Atrial flutter (Cardiac disorders) | 4
Ventricular fibrillation (Cardiac disorders) | 4
Atrioventricular block complete (Cardiac disorders) | 3
Mitral valve incompetence (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 3
Aortic valve incompetence (Cardiac disorders) | 2
Atrioventricular block second degree (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 2
Cardiac tamponade (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 2
Atrial thrombosis (Cardiac disorders) | 2
Cardiac valve disease (Cardiac disorders) | 2
Stress cardiomyopathy (Cardiac disorders) | 2
Aortic valve stenosis (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Nodal arrhythmia (Cardiac disorders) | 1
Pericardial haemorrhage (Cardiac disorders) | 1
Prinzmetal angina (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Tachycardia paroxysmal (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Intracardiac thrombus (Cardiac disorders) | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Arterial occlusive disease (Vascular disorders) | 3
Deep vein thrombosis (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 2
Aortic aneurysm (Vascular disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Peripheral artery aneurysm (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 15
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 12
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 6
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6
Ileus (Gastrointestinal disorders) | 6
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5
Large intestine polyp (Gastrointestinal disorders) | 5
Colitis ischaemic (Gastrointestinal disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 3
Melaena (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Inguinal hernia (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Oesophageal dysplasia (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 4
Cholangitis acute (Hepatobiliary disorders) | 3
Drug-induced liver injury (Hepatobiliary disorders) | 3
Cholecystitis acute (Hepatobiliary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Biliary cirrhosis primary (Hepatobiliary disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Gallbladder polyp (Hepatobiliary disorders) | 1
Hepatic mass (Hepatobiliary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 4
Renal impairment (Renal and urinary disorders) | 4
Acute kidney injury (Renal and urinary disorders) | 2
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal infarct (Renal and urinary disorders) | 1
Renal tubular necrosis (Renal and urinary disorders) | 1
Urogenital haemorrhage (Renal and urinary disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 1
Renal mass (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 1
Death (General disorders) | 11
Sudden death (General disorders) | 3
Multiple organ dysfunction syndrome (General disorders) | 3
Asthenia (General disorders) | 1
Condition aggravated (General disorders) | 1
Drowning (General disorders) | 1
Drug interaction (General disorders) | 1
Generalised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Disuse syndrome (General disorders) | 1
Occult blood positive (Investigations) | 2
Activated partial thromboplastin time prolonged (Investigations) | 1
White blood cell count increased (Investigations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 12
Fall (Injury, poisoning and procedural complications) | 8
Femoral neck fracture (Injury, poisoning and procedural complications) | 4
Contusion (Injury, poisoning and procedural complications) | 3
Road traffic accident (Injury, poisoning and procedural complications) | 2
Accident (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Brain contusion (Injury, poisoning and procedural complications) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Varicose vein operation (Surgical and medical procedures) | 1
Cancer surgery (Surgical and medical procedures) | 1
Large intestinal polypectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With NVAF (N=6443)
Dyspepsia (Gastrointestinal disorders) | 408

LIMITATIONS AND CAVEATS:
The study was conducted in an unblinded manner and without controls. The explanatory power of the study results was limited and the study results should be interpreted with the necessary caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No